CLINICAL TRIAL: NCT04682275
Title: Gender Differences in Periodontal Status of Depressive and Non-Depressive Individuals
Brief Title: Effect of Gender on Depression and Periodontal Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Uçan Yarkaç, Principal Investigator, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NecmettinCT
Record Dates: First submitted 2020-12-06; First posted 2020-12-23 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Periodontal Diseases; Depression; Gender; Gingival Diseases
Keywords: periodontal diseases; depression; gender; gingival diseases
MeSH Terms: conditions — Periodontal Diseases; Depression; Coitus; Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Female Group (Other): Females with periodontal disease (71 subjects with gingivitis, 100 subjects with periodontitis)
  Interventions: Other: Psychological measurements
- Male Group (No Intervention): males with periodontal disease (72 subjects with gingivitis, 96 subjects with periodontitis)

INTERVENTIONS:
Other: Psychological measurements — A questionnaire test (Beck depression Inventory) for depression was performed.
  Arms: Female Group

SUMMARY:
There is a relationship between depression and periodontal disease. This relationship may be double-sided. A psychological state such as anxiety, depression, body image, and self-esteem may be affected from the symptoms of periodontal disease.

DETAILED DESCRIPTION:
Background: Depression is a multifactorial disease characterized by a variety of symptoms. Individuals with psychiatric disorders seem to be more prone to periodontitis. However periodontal disease and depression can be considered bidirectional risk factors. Periodontal diseases can also be an effect on depression. The purpose of the present study was to evaluate the gender-related differences in the relationship between periodontal diseases and depression in male and female adults.

Material and methods: The study population consisted of 339 subjects. Two groups were formed from these patients: 171 females with periodontal disease (71 subjects with gingivitis, 100 subjects with periodontitis); 168 males with periodontal disease (72 subjects with gingivitis, 96 subjects with periodontitis). Clinical periodontal and psychological measures were performed on females and males group.

ELIGIBILITY:
Inclusion Criteria:

* the presence of periodontal diseases

Exclusion Criteria:

* the presence of any systemic disease other than depression
* smoking and alcohol consumption
* the use of any drugs (antidepressants, anti-inflammatory, and antimicrobial medicaments, and hormonal supplements) that affect the periodontal condition
* have received any periodontal treatment in the last six months
* hormonal condition such as pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2017-03-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Depression level | Baseline
  The differences in depression level between females and males. Depression level was determined using the Beck Depression Inventory.
  Beck Depression Inventory (BDI) consists of 21 items. Each of the 21 statements is scored from 0 to 3. The total score allows the classification of depression severity. Scores less than 10 indicates lack of the depression. The scores between10-16 indicate minimum depression, the scores between17-29 indicate moderate depression, scores greater than 30 indicate severe depression.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline
  Probing pocket depth (PPD) was measured for determining the severity of the disease and clinical outcome. High probing pocket depth shows more severe periodontal disease.
Gingival index | Baseline
  The differences in gingival index scores between females and males. The gingival index was recorded for determining and classifying gingival status. The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding.
Plaque index | Baseline
  The differences in plaque index scores between females and males. Plaque index (PI) was recorded for determining and classifying oral hygiene status. The Plaque Index (GI) scores each site on a 0 to 3 scale with 0 being no plaque in the gingival area and 3 abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
Bleeding on probing | Baseline
  The differences in bleeding on probing scores between females and males. Bleeding on probing (BOP) has been used to diagnose the presence of periodontal diseases, and it is a reliable indicator of gingival inflammation. It is useful in providing either positive predictive values or negative predictive values that illustrate disease progression. A positive predictive value indicates the percentage of people who both exhibit BOP and are correctly diagnosed with progressive periodontal diseases. A negative predictive value indicates the percentage of people whose BOP test results show no bleeding and no active disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ucan Yarkac, 1, Principal Investigator — Necmettin Erbakan University; Ozge Gokturk, 1, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No